CLINICAL TRIAL: NCT05746052
Title: Microneedling Versus Punch Elevation With Microneedling in Treatment of Atrophic Acne Scars: Comparative Study
Brief Title: Punch Elevation and Microneedling in Treatment of Atrophic Acne Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud Mohamed Mahmoud, MSc researcher, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSc/AZ.AST./DVA21/12/194/4/202
Record Dates: First submitted 2023-02-17; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Acne Scars

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- atrophic acne scar in face (Other)
  Interventions: Procedure: Punch insturment

INTERVENTIONS:
Procedure: Punch insturment — surgical and dermatological tool used mainly for skin biopsy and therapeutic skin disorders

SUMMARY:
The ultimate goal of this study was to compare punch elevation and micro needling with PRP versus micro needling and PRP only in treatment of post acne scars, in an attempt to achieve better management of such condition.

This is a prospective study that was carried out on 15 patients (their ages ranged from 19 to 32 years with a mean of 23 years. They are 6 males and 7 females, 7 patients were of skin photo type III, and 10 were rural residents), they presented with post acne facial scars, and attending the Dermatology and Andrology outpatient clinic of Al-Azhar University Hospital in (Assiut), between April 2021 and March 2022. Left side of face of the lesion of each patient will be treated by punch elevation two weeks before microneeedling with platlets rich plasma (PRP),the right side will be treated by microneedling with (PRP) only from the start, three sessions of microneedling will be done with 4 weeks interval.

Each patient had punch elevation for scars in left side at first session then dressing removed after 7 days after three weeks all patents received treatment on both sides of the face by micro needling with PRP.

During each session, topical anesthesia was applied over the area of interest on face and removed after 20 mints. Patients were placed in supine position with head stable, the skin was stretched and micro needling was carried out in vertical, horizontal and both diagonal directions for about 4-5 times. PRP (2 ml) were applied on the face. A total of three sessions of microneedling were performed at monthly intervals.

Follow-up of the patients was done before and after treatment by clinical examination and photography by comparing the photographs before and after therapy; Evolution of clinical response included extent of improvement and possible adverse effects including bleeding, and erythema. And PIH Clinical photos of the lesions had been taken before the first session and one month after the last session and assessed clinically to grade the severity of scarring proposed by Goodman and Baron's quantitative scale for acne scars at the baseline and the end of study. Patients' satisfaction had been done by using a quartile grading system (1 poorly satisfied, 2 satisfied or 3 very satisfied).

As regard efficacy of the procedures, we found significant improvement of atrophic acne scars, with significant reduction in number of acne scars as well as significant reduction in goodman score after treatment by punch elevation and micro needling with PRP, most of patients were satisfied after treatment, the side treated with punch elevation have statistically significant reduction in the number of the scar when compared to the right side.

ELIGIBILITY:
Inclusion Criteria:

Patients of both genders. Patients with Ice pick and box scars of any duration. Co-operative patients and patients are willing for the procedure. Patients of age 18 - 40 years

Exclusion Criteria:

Presence of active acne lesions. Patients with active infection at the local site or recurrent herpes. Patients with history of bleeding disorders or anticoagulant medications Patients with keloid scarring or hypertrophic scar. patients with recurrent herpes simplex infection

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
change in acne scars | 4 weeks following end of treatment
  Goodman and Baron's quantitative acne scar grading system

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine AlAzhar University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No